CLINICAL TRIAL: NCT01301209
Title: Prospective Observational Study of Recto-Anal-Repair in the Treatment Haemorrhoidal Disease Stage III/IV
Brief Title: Recto-Anal-Repair in the Treatment of Advanced Haemorrhoidal Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Sebastian Roka/MD, Dept. of General Surgery, Medical University Vienna
Other Study IDs: 078/2006
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2006-06

CONDITIONS: Haemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment: patients undergoing treatment

SUMMARY:
Prospective observational study to evaluate the impact of Recto-Anal-Repair (a technique of ultrasound guided haemorrhoidal ligation) in the treatment of stage III/IV haemorrhoidal disease.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV hemorrhoidal disease (Appendix A)
* Patient age 18-80 years old
* Patient fit for general or local anesthesia
* No prior surgical treatment for hemorrhoidal disease
* No prior surgical treatment for anorectal sepsis
* Signed informed consent

Exclusion Criteria:

* Stage I or II hemorrhoidal disease (Appendix A)
* Patient unfit for surgery
* Clotting disorders
* Anal or colorectal malignancy
* Secondary hemorrhoidal disease
* Pregnancy
* Unwilling or unable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with haemorrhoids stage III/IV
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Roka, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Dept. of Surgery, Medical University Vienna, Vienna, Vienna, Austria